CLINICAL TRIAL: NCT04078776
Title: Systemic and White Adipose Tissue Inflammatory Profile in Lean Versus Obese Individuals
Status: Completed | Type: Observational
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Dr Oonagh Markey, Vice-Chancellor's Research Fellow, Loughborough University
Other Study IDs: R19-P144
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Inflammation; Obesity; Inflammatory Response; Cardiovascular Risk Factor
MeSH Terms: conditions — Inflammation; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean Individuals: waist circumference ≤94 cm (men) and 80 cm (women) and BMI ≥ 21.0 kg/m2
  Interventions: Other: No intervention
- Obese Individuals: waist circumference ≥102cm (men) and 88 cm (women) and BMI ≥ 30.0kg/m2
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention in this study

SUMMARY:
This study will compare the systemic and white adipose tissue inflammatory profile of individuals who are classified as lean and obese. Blood and white adipose tissue samples will be collected in the fasted state to assess inflammatory status.

There is evidence to suggest that markers of inflammation in the blood and white adipose tissue increase with increasing levels of obesity. However, the white adipose tissue total protein content and phosphorylation of proteins involved in inflammatory pathways has not previously been compared between lean and obese individuals.

The investigators hypothesise that obese individuals will have increased levels of inflammation in the blood and white adipose tissue, compared to their lean counterparts.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Waist circumference/BMI criteria:

  * Lean participants: waist circumference ≤94 cm (men) and 80 cm (women) and BMI ≥ 21.0 kg/m2 or
  * Obese participants: waist circumference ≥102 cm (men) and 88 cm (women) and BMI ≥ 30.0kg/m2
* Recreationally active (> 3 x 30 min moderate exercise per week)
* Blood pressure systolic blood pressure <160 mmHg and diastolic blood pressure <100 mmHg

Exclusion Criteria:

* Smoker (including vaping)
* Cardiometabolic or inflammatory disease (e.g. heart disease, high blood pressure, type 2 diabetes)
* Taking medication or nutritional supplements (e.g. fish oil/prebiotics) known to interfere with study outcomes (including inflammation, immune function or lipid/carbohydrate metabolism) or prescribed antibiotics within the last 3 months
* Unstable weight history (≥ 3kg loss or gain in previous 3 months)
* An allergy to lidocaine (determined by the Schools standard health questionnaire)
* Parallel participation in another intervention study
* Women who are pregnant or lactating
* Any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a metabolic study
* Alcohol consumption >28 units per week for a man or >21 units per week for a woman

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Apparently healthy, recreationally active adults.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Protein expression (content and phosphorylation) of key markers of metabolic inflammation in white adipose tissue (for example assessment of Nuclear factor kappa B (NFKB) total protein and phosphorylation by western blot analysis) | Cross-sectional (all outcome measures will be collected within a 2 week period)
  This will be assessed following the collection of fasted white adipose tissue samples

SECONDARY OUTCOMES:
Systemic Markers of Inflammation (for example C-reactive protein and interleukin 6 concentrations, determined by spectrophotometric assay/ ELISA) | Cross-sectional (all outcome measures will be collected within a 2 week period)
  This will be assessed following the collection of fasted white adipose tissue
Gene expression of key markers of metabolic inflammation in white adipose tissue | Cross-sectional (all outcome measures will be collected within a 2 week period)
  This will be assessed following the collection of fasted white adipose tissue
Characterisation of immune cell populations (monocyte subsets) from peripheral blood mononuclear cells (measured using flow cytometry analysis) | Cross-sectional (all outcome measures will be collected within a 2 week period)
  This will be assessed following the collection of fasted blood samples
Habitual Dietary Intake | Cross-sectional (all outcome measures will be collected within a 2 week period)
  This will be assessed following the collection of a 4 day weighed food diary
Physical Activity | Cross-sectional (all outcome measures will be collected within a 2 week period)
  Assessed using Actigraph accelerometers over a 4 day period
Fasting Serum Markers of Insulin Resistance (for example insulin and glucose concentrations, determined using an ELISA/ spectrophotometric assay) | Cross-sectional (all outcome measures will be collected within a 2 week period)
  This will be assessed following the collection of fasted blood samples
Fasting Serum Lipid Profile (for example total cholesterol, HDL cholesterol and triacylglycerol concentrations, measured using a spectrophotometric assay) | Cross-sectional (all outcome measures will be collected within a 2 week period)
  This will be assessed following the collection of fasted blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Oonagh Markey, BSc, PhD, Principal Investigator — Vice-Chancellor's Research Fellow, Loughborough University
Locations (1):
- Loughborough University, Loughborough, United Kingdom